CLINICAL TRIAL: NCT06444945
Title: Effects of Mulligan Mobilization With Movement as Compared to Kaltenborn Joint Mobilization in the Management of Knee Osteoarthritis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/13
Record Dates: First submitted 2024-05-27; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Transcutaneous Electric Nerve Stimulation; Movement; Resistance Training

STUDY DESIGN:
Intervention Model Description: Parallel designed randomized control trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan MWM group (Experimental): Group A receiving Mulligan MWM joint mobilization
  Interventions: Device: Heating pad; Device: Transcutaneous electrical nerve stimulation(TENS); Procedure: Mulligan mobilization with movement (MWM); Procedure: Resistance Training exercise
- Kaltenborn mobilization group (Experimental): Group B receiving Kaltenborn Joint mobilization
  Interventions: Device: Heating pad; Device: Transcutaneous electrical nerve stimulation(TENS); Procedure: Kaltenborn joint mobilization; Procedure: Resistance Training exercise

INTERVENTIONS:
Device: Heating pad — Heating pad will be used for heating purpose.
Device: Transcutaneous electrical nerve stimulation(TENS) — TENS is used for symptomatic pain relief
Procedure: Mulligan mobilization with movement (MWM) — It provides short term pain relief and to restore pain-free, functional movements by achieving full range at the joint
  Arms: Mulligan MWM group
Procedure: Kaltenborn joint mobilization — The purpose of joint mobilization is to restore normal, painless joint function. In restricted joints, this involves the restoration of joint play to normalize the roll-gliding that is essential to active movement.
  Arms: Kaltenborn mobilization group
Procedure: Resistance Training exercise — Resistance training increases muscle strength by making your muscles work against a weight or force.

SUMMARY:
This study is a randomised controlled trial and the purpose of this study is to determine the Effects of Mulligan mobilization with movement as compared to Kaltenborn joint mobilization in the management of knee osteoarthritis." To determine the effects of Mulligan MWM as compared to Kaltenborn joint mobilization in terms of pain, function, range of motion and gait in persons with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 40-70 years (Osama et al, 2022)
* Having KOA history of no less than 3 months
* Knee pain less than 8/10 on numeric pain rating scale (NPRS).
* Radiological evidence of grade III or less on Kellgren classification
* Patients referred from rehab department

Exclusion Criteria:

* Those with signs of serious pathology, such as malignancy, inflammatory disorder or infection.
* History of trauma or fractures in lower extremity.
* Signs of lumbar radiculopathy or myelopathy.
* History of knee surgery or replacement.
* Receiving intra-articular steroid therapy in the preceding two months.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-10 (Estimated); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
knee pain | 2 weeks
  knee pain will be measured using visual analogue scale (VAS) from 0-100mm.A higher score on VAS indicated greater pain.
Functional disability | 2 weeks
  knee functional disability will be assessed using Knee Osteoarthritis and Outcome Score(KOOS) with a score ranging from 0-100. A lower score on KOOS signifies greater functional disability
Knee range of motion | 2 weeks
  knee range of motion will be measured using a goniometer. A higher ROM signifies positive outcome.
Stride length | 2 weeks
  Gait analysis will be done to analyze stride length. A greater stride length signifies positive outcome and prognosis.
Gait velocity | 2 weeks
  Gait analysis will be done to analyze gait velocity. A greater gait velocity signifies positive outcome and prognosis.
Isometeric Muscle Strength | 2 weeks
  Isometeric Muscle Strength will be quantified using dynamometer. A higher score on dynamometer signifies greater muscle strength and good prognosis.
Walking related performance fatigability | 2 weeks
  walking related performance fatigability will be measured using 6 minute walk test. Greater fatigibility indicates poorer outcome.
Functional Capacity | 2 weeks
  5 repetition sit to stand test will be used to determine knee related functional capacity which will be quantified in terms of time. A smaller time will denote greater functional capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Shanza Fatima, DPT, Principal Investigator — Foundation University Islamabad; Muhammad Osama, PHD*, Principal Investigator — Foundation University Islamabad
Locations (1):
- Foundation University Islamabad, Islamabad, Pakistan